CLINICAL TRIAL: NCT03195595
Title: Minimal Invasive Mitral Valve Replacement Versus Conventional Median Sternotomy Approach
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Elhussein Mohamed Abdelmottaleb, Resident doctor at cardiothoracic surgery, Assiut University
Other Study IDs: 17100176
Record Dates: First submitted 2017-06-05; First posted 2017-06-22 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Mitral Valve Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mitral valve replacement: patients whom underwent Mitral valve replacement through minimal invasive incision
  Interventions: Device: mitral valve replacement; Device: conventional mitral valve replacement
- conventional mitral valve replacement: patients whom underwent Mitral valve replacement through conventional sternotomy

INTERVENTIONS:
Device: mitral valve replacement — early postoperative outcome regarding pain in minimal invasive technique
  Groups: mitral valve replacement
Device: conventional mitral valve replacement — early postoperative outcome regarding pain in conventional median sternotomy
  Groups: mitral valve replacement

SUMMARY:
This is retrospective study that will be done in Cardiothoracic surgery department in Assuit university hospitals for one year duration aiming to compare minimal invasive technique to conventional median sternotomy for mitral valve surgery regarding early postoperative outcomes and pain

DETAILED DESCRIPTION:
This is retrospective study that will be done in Cardiothoracic surgery department in Assuit university hospitals for one year duration and the study tools will be:

Part I (Demographic data):

* Age, Gender, Weight, Height ,Smoke history

Part II (Preoperative data):

* Medical history, Clinical assessment, Preoperative investigation

Part III (Intraoperative data):

* Surgical time, and Ischemic time

Part IV (Postoperative data):

* Early ambulation, ICU stay, length of ventilation, using of analgesic drugs, post op bleeding, deaths

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with mitral valve disease indicated for valve surgery

Exclusion Criteria:

* Double valve disease or other valve disease
* Mitral or aortic valve disease associated with ischemic heart disease
* Mitral or aortic valve disease associated with congenital heart disease
* Patients subjected to prior heart surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It includes groups of population above age of 18 with symptomatic mitral valve disease indicated for valve surgery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluating of postoperative pain by using numerical rating scales (NRS) | one year
  its a score result from gathered information from the patient

SECONDARY OUTCOMES:
Evaluating early postoperative outcome | one year
  e.g., bleeding

CONTACTS AND LOCATIONS:
Overall Officials: mohamed A nady, lecturer, Study Director — Assuit university hospital
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No